CLINICAL TRIAL: NCT06050941
Title: A Multi-center Prospective Single Arm Clinical Study of Reduced Intensive 3 + 5 Idarubicin and Cytarabine Chemotherapy Plus Venetoclax as First-line Treatment for Adults With Acute Myeloid Leukaemia and High-risk Myelodysplastic Syndrome
Brief Title: Reduced Intensive Idarubicin and Cytarabine Plus Venetoclax as First-line Treatment for Adults AML and MDS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Weiyan Zheng, Clinical Professor, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230413IAVEN
Record Dates: First submitted 2023-04-13; First posted 2023-09-22 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-04

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Idarubicin; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Reduced intensive of 3 + 5 Idarubicin and Cytarabine plus Venetoclax as induction therapy
  Interventions: Drug: idarubicin; Drug: Cytarabine

INTERVENTIONS:
Drug: idarubicin — Idarubicin 6mg/m2 d5-7
  Other Names: Idamycin; Demethoxydaunorubicin
Drug: Cytarabine — Cytarabine 60mg/m2 d5-9
  Other Names: Cytosar; Cytosine arabinoside

SUMMARY:
Reduced intensive 3 + 5 idarubicin and cytarabine chemotherapy plus venetoclax as first-line treatment for adults with acute myeloid leukaemia and high-risk myelodysplastic syndrome

DETAILED DESCRIPTION:
Multiple clinical trials about chemotherapy plus venetoclax in primary diagnosed AML or relapsed/refractly AML were ongoing to attempt the facility of the combination. Zu et al demostrated that full dose of 3 + 7 daunorubicin and cytarabine chemotherapy plus 8 days escalated venetoclax acheived 91% of CR/CRi with 97% 1-year overall survival and 72% 1-year event-free survival. In this trial , we try to reduced the intensive of 3 + 5 idarubicin and cytarabine chemotherapy, but prolong venetoclax to two weeks in the induction therapy in adults AML/MDS. We expect to increase the induced remission rate by extending the dosage of targeted drug venetoclax, and minimize the side effects by reducing the dose of 3 + 7 induction chemotherapy, so as to achieve the goal of high efficiency and low toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-60 years
2. had a confirmed diagnosis of previously untreated de novo acute myeloid leukaemia or high risk myelodysplastic syndrome by bone marrow examination according to the criteria presented by WHO.
3. Eastern Cooperative Oncology Group performance status of 0-2.
4. adequate renal and hepatic function (appendix 2 p 45), and left ventricular ejection fraction of at least 45% by echocardiography.

Exclusion Criteria:

1. younger than 18 years old, or older than 60 years old.
2. Diagnosed as acute promyelocytic leukaemia.
3. Pretreated with anthracycline.
4. CNS involvement.
5. Positive for HIV, hepatitis B virus, or hepatitis C virus.
6. New York Heart Association cardiovascular disability status higher than grade 2 (grade 2 is defined as cardiac disorder that is asymptomatic at rest, but ordinary physical activity might result in fatigue, palpitations, dyspnoea, or angina), chronic respiratory diseases requiring continuous supplementary oxygen, inability to take oral medication or malabsorption syndrome
7. Uncontrollable systemic infection (viral, bacterial, or fungal),
8. Inability to sign the informed consent form.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-02 (Estimated); Primary Completion 2026-04-02 (Estimated); Study Completion 2027-04-02 (Estimated)

PRIMARY OUTCOMES:
CR | Week 6
  assessment of the composite complete remission rate (CR=CR+CRi)

SECONDARY OUTCOMES:
MRD | Week 6
  assessment of bone marrow measurable residual disease by flow cytometry
EFS | 2 years
  Evaluate the event-free survival
OS | 2 years
  Evaluated the overall survival
adverse events | at any time
  Monitor of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Weiyan Zheng, MD, Principal Investigator — Zhejiang University